CLINICAL TRIAL: NCT05788068
Title: Efficacy and Neuroimaging Mechanisms of Smoking Cessation in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Yanhui Liao, Deputy Chief Physician, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220061
Record Dates: First submitted 2023-02-22; First posted 2023-03-28 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Cigarette Smoking; Psychological Interventions; Smoking Cessation
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants in the intervention group will receive CBT-based digital smoking cessation intervention. The intervention is a set of smoking cessation methods based on the theoretical study of cognitive behavioral therapy for smoking cessation, and its effectiveness has been confirmed through our large sample of randomized controlled studies. This study plans to intervene smokers for 4 weeks after the start of smoking cessation.
  Interventions: Behavioral: Cognitive behavior therapy

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — Participants will receive CBT intervention for smoking cessation via "wechat"-based mini-program developed by a professional team.

SUMMARY:
This proposed project is to assess the efficacy of CBT-based digital smoking cessation interventions in China, as well as explore its neuroimaging mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Use cigarettes for no less than 1 year, and use cigarettes ≥ 10 per day
2. Nicotine dependence (FTCD ≥ 3)
3. Willing to make an attempt to quit smoking in the next month, and have not quit smoking in the past 3 months, and .
4. No other addictions except nicotine
5. Education level of junior high school or above
6. Age between 18 to 45 years old
7. Right-handed
8. No contraindication of MRI scanning
9. Willing to provide informed consent to participate in the study.

Exclusion Criteria:

1. Patients who are receiving medication
2. Previous and current mental disorders,and/or mental disorders in line with DSM-5 diagnostic criteria in two departments and three generations.
3. Brain organic disease, brain injury history, coma history
4. Serious physical disease, endocrine disease history, abnormal blood picture, heart, liver and kidney function after examination
5. Pregnant and lactating women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Biochemically Validated Continuously Abstinence | 4 weeks
  Biochemical validation of 4-week continuous smoking abstinence by urine cotinine test.
Brain Structural Characteristics | 4 weeks
  Differences of brain structure between successful and unsuccessful smokers after intervention, which will be measured by white matter volume, gray matter volume, cortical thickness, and surface area.
Brain Functional activity | 4 weeks
  Differences of whole brain function activity between successful and unsuccessful smokers after intervention, which will be measured by ReHo, ALFF, fALFF, and functional connectivity (FC)

SECONDARY OUTCOMES:
Self-reported 7-day Point Abstinence | 4 weeks
  Self-reported 7-day point-prevalence abstinence at week 1, 4, 8, 12, 16, 20 and 26 after quit date.
Self-reported Continuous Abstinence | 4 weeks
  Self-reported continuous smoking abstinence rate at weeks 4, 8, 12, 16, 20, and 26 after the quit date.

OTHER OUTCOMES:
Smoking Reduction and Participation | 4 weeks
  Reductions in number of cigarettes smoked per day and rates of participation in and completion of smoking-cessation programs.

CONTACTS AND LOCATIONS:
Locations (1):
- Yanhui Liao, Hanzhou, Zhejiang, China